CLINICAL TRIAL: NCT03347448
Title: Beijing University of Chinese Medicine
Brief Title: Multidimensional Cross-sectional Study on Skin Health Based on TCM Constitution - Psychology - Skin Model
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Beijing University of Chinese Medicine (Other)
Responsible Party: Principal Investigator, Tuya Bao, Professor, Beijing University of Chinese Medicine
Other Study IDs: BeijingUCMPS
Record Dates: First submitted 2017-10-31; First posted 2017-11-20 (Actual); Last update posted 2017-11-20 (Actual); Status verified 2017-11

CONDITIONS: Psychology; Skin
Keywords: Psychology; Skin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

SUMMARY:
This survey was designed as a cross-section study investigation, after the selection,the invesgators would adopt the methods of randomly drawing for 100 Beijing female citizens to process: questionnaire survey about the skin health, infrared thermal imaging on facing area, VISIA skin testing and Germany CK company skin testing etc. for integrated evaluation of skin health.

This survey was designed as a cross-section study investigation, after the selection,the invesgators would adopt the methods of randomly drawing for 100 Beijing female citizens to process: questionnaire survey about the skin health, infrared thermal imaging on facing area, VISIA skin testing and Germany CK company skin testing etc. for integrated evaluation of skin health. Analyzing the constitution of volunteers and combining the test related to depression and anxious, psychology health evaluated the healthy states. Base on the data collected processed the statistic analyzing, comprehensive assessment the impact factor of skin health for establishing the Constitution-Psychology-Skin model and though this model to evaluate and forecast the skin health problem.

DETAILED DESCRIPTION:
This survey the invesgators designed as a cross-section study investigation, after the selection,the invesgators would adopt the methods of randomly drawing for 100 Beijing female citizens to process: questionnaire survey about the skin health, infrared thermal imaging on facing area, VISIA skin testing and Germany CK company skin testing etc. for integrated evaluation of skin health.

This survey was designed as a cross-section study investigation, after the selection,the invesgators would adopt the methods of randomly drawing for 100 Beijing female citizens to process: questionnaire survey about the skin health, infrared thermal imaging on facing area, VISIA skin testing and Germany CK company skin testing etc. for integrated evaluation of skin health. Analyzing the constitution of volunteers and combining the test related to depression and anxious, psychology health evaluated the healthy states. Base on the data collected processed the statistic analyzing, comprehensive assessment the impact factor of skin health for establishing the Constitution-Psychology-Skin model and though this model to evaluate and forecast the skin health problem.

Standards of included:

1. Female,
2. Ages between 18 or above, 55 or below,
3. Informed consent, voluntary.

Standards of excluded:

1. Taking part in other surveys before the starting of this survey within 2 months,
2. Obviously disturbance of consciousness,
3. Suffering from endocrine systemic disease, mental disease or other severe systemic disease,
4. Pregnant or lactation period,
5. Researchers consider that would occur harmful toward volunteers or would affect the aims and the explanation of the results.

The volunteers must require all the above standards would conform to the selection.

Standards of retreat from this survey:

1. Poor compliance, could not complete all the tests,
2. Occur any special physiological and pathological changes which not suitable for funder process.

ELIGIBILITY:
Inclusion Criteria:

1. Female,
2. Ages between 18 or above, 55 or below,
3. Informed consent, voluntary.

Exclusion Criteria:

Exclusion Criteria:

1. Taking part in other surveys before the starting of this survey within 2 months,
2. Obviously disturbance of consciousness,
3. Suffering from endocrine systemic disease, mental disease or other severe systemic disease,
4. Pregnant or lactation period,
5. Researchers consider that would occur harmful toward volunteers or would affect the aims and the explanation of the results.

Ages: 15 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Female,Ages between 18 or above, 55 or below,Informed consent, voluntary.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-11-18 (Estimated); Primary Completion 2018-02-15 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
PHQ-9 | 1 year
  PRIME-MD diagnostic instrument for common mental disorders.
PSQI | 1 year
  Despite the prevalence of sleep complaints among psychiatric patients, few questionnaires have been specifically designed to measure sleep quality in clinical populations.
SCL-90 | 1 year
  SCL-90 relatively brief self-report psychometric instrument (questionnaire) published by the Clinical Assessment division of the Pearson Assessment & Information group. It is designed to evaluate a broad range of psychological problems and symptoms of psychopathology. It is also used in measuring the progress and outcome of psychiatric and psychological treatments or for research purposes.
SAS | 1 year
  The SAS is a 20-item self-report assessment device built to measure anxiety levels, based on scoring in 4 groups of manifestations: cognitive, autonomic, motor and central nervous system symptoms. Answering the statements a person should indicate how much each statement applies to him or her within a period of one or two weeks prior to taking the test.
Infrared thermal imaging | 1 year
  To measure the condition of the skin.
VISIA skin testing | 1 year
  To measure the condition of the skin.
Moisture content | 1 year
  To measure the condition of the skin.
Haematochrome test | 1 year
  To measure the condition of the skin.
Elasticity Test of Skin | 1 year
  To measure the condition of the skin.
Skin Sebum Test | 1 year
  To measure the condition of the skin.
Glossiness of Skin | 1 year
  To measure the condition of the skin.
Neuronal Sensitivity | 1 year
  To measure the condition of the skin.
Melanin Test | 1 year
  To measure the condition of the skin.
Chroma of Skin | 1 year
  To measure the condition of the skin.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Wolf R, Wolf D, Tamir A, Politi Y. Melasma: a mask of stress. Br J Dermatol. 1991 Aug;125(2):192-3. doi: 10.1111/j.1365-2133.1991.tb06075.x. No abstract available. PMID 1911305